CLINICAL TRIAL: NCT04484311
Title: Multi-center Survey on Non-curative ESDs: Assessing the Rates and Risk Factors for Residual Neoplasia
Brief Title: Non-curative ESDs: Assessing the Rates and Risk Factors for Residual Neoplasia
Acronym: NC-ESD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Other Study IDs: Non-Curative ESDs Registry
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-07

CONDITIONS: Gastric Neoplasm; Esophageal Neoplasms; Colorectal Neoplasms
Keywords: Endoscopic therapy; Endoscopic submucosal dissection
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Short and long outcomes of ESD are well described, particularly in Eastern series. However, the outcome of non-curative ESDs is scarcely reported in the west (particularly among non-gastric or submucosal lesions). Therefore, the aim of this project is to describe the European experience with non-curative ESDs, analysing all the consecutive ESDs performed in several reference centers, assessing the presence of residual lesion in the endoscopic follow-up or in the surgical specimen.

ELIGIBILITY:
Inclusion Criteria:

* All patients submitted to ESD due to neoplastic lesions of the gastrointestinal tract

Exclusion Criteria:

* Patients without endoscopic follow-up or surgery will be excluded from the analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients submitted to ESD due to neoplastic lesions of the gastrointestinal tract.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Residual neoplasia | 2010-2020
  Presence of residual neoplasia after non-curative ESD

CONTACTS AND LOCATIONS:
Overall Officials: João Santos-Antunes, Principal Investigator — Gastrointestinal Department, Centro Hospitalar S. João, Porto, Portugal; Guilherme Macedo, MD, PhD, Study Director — Gastrointestinal Department, Centro Hospitalar S. João, Porto, Portugal
Locations (1):
- Hospital S. João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morais R, Libanio D, Dinis Ribeiro M, Ferreira A, Barreiro P, Bourke MJ, Gupta S, Amaro P, Kuttner Magalhaes R, Cecinato P, Boal Carvalho P, Pinho R, Rodriguez de Santiago E, Sferrazza S, Lemmers A, Figueiredo M, Pioche M, Gallego F, Albeniz E, Ramos Zabala F, Uchima H, Berr F, Wagner A, Marques M, Pimentel-Nunes P, Goncalves M, Mascarenhas A, Soares EG, Xavier S, Faria-Ramos I, Sousa-Pinto B, Gullo I, Carneiro F, Macedo G, Santos-Antunes J. Predicting residual neoplasia after a non-curative gastric ESD: validation and modification of the eCura system in the Western setting: the W-eCura score. Gut. 2023 Dec 7;73(1):105-117. doi: 10.1136/gutjnl-2023-330804. PMID 37666656
- [Derived] Santos-Antunes J, Pioche M, Ramos-Zabala F, Cecinato P, Gallego Rojo FJ, Barreiro P, Felix C, Sferrazza S, Berr F, Wagner A, Lemmers A, Figueiredo Ferreira M, Albeniz E, Uchima H, Kuttner-Magalhaes R, Fernandes C, Morais R, Gupta S, Martinho-Dias D, Rios E, Faria-Ramos I, Marques M, Bourke MJ, Macedo G. Risk of residual neoplasia after a noncurative colorectal endoscopic submucosal dissection for malignant lesions: a multinational study. Endoscopy. 2023 Mar;55(3):235-244. doi: 10.1055/a-1906-8000. Epub 2022 Jul 21. PMID 35863354